CLINICAL TRIAL: NCT03492931
Title: A Multi-centre, Phase I, Open-label, Single-dose Study to Investigate Pharmacokinetics (PK) of Ticagrelor in Infants and Toddlers, Aged 0 to Less Than 24 Months, With Sickle Cell Disease (HESTIA4)
Brief Title: PK Study of Ticagrelor in Children Aged Less Than 24 Months, With Sickle Cell Disease (HESTIA4)
Acronym: HESTIA4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D5136C00010
Record Dates: First submitted 2018-03-16; First posted 2018-04-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Sickle Cell Disease
Keywords: Hb SS disease, Hb S Beta 0 Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Ticagrelor

STUDY DESIGN:
Masking Description: Study has an Open-Label design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Single dose of ticagrelor based on age
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Patients will receive a single dose of ticagrelor
  Other Names: AR-C124910XX is an active metabolite of ticagrelor given orally in a single dose. It will be measured, but it won't be given directly to subjects.

SUMMARY:
The purpose of this Phase I study is to investigate the pharmacokinetic properties of ticagrelor in pediatric patients from 0 to less than 24 months with sickle cell disease.

Ticagrelor dose level adjustment will require a Protocol amendment and regulatory approval.

DETAILED DESCRIPTION:
Study design This Phase I paediatric study (in patients aged 0 to <24 months) with ticagrelor is planned to be a multi-centre, open-label, single dose study.

Primary Objective:

To determine the PK properties of ticagrelor after a single oral dose

Secondary Objectives:

To determine the PK properties of the active metabolite (AR-C124910XX) after a single oral dose To assess the acceptability and the palatability of a single oral dose of ticagrelor

Safety Objective:

To assess safety and tolerability of a single oral dose of ticagrelor

Duration of treatment At least 20 eligible patients will receive a single open label oral dose of ticagrelor on Day 1.

Statistical methods A population PK analysis approach will be used to determine the PK parameters of ticagrelor and its metabolite AR-C124910XX in paediatric patients aged 0 to <24 months eg, CL/F (oral clearance) (only for ticagrelor) and AUC.

The PK will also be described by presenting the observed plasma concentrations of Ticagrelor and its active metabolite for all individuals, as well as corresponding descriptive statistics.

No statistical comparisons are planned for the primary or secondary objectives, which will be summarised descriptively

ELIGIBILITY:
Inclusion Criteria:

1. Paediatric patients aged <24 months, diagnosed with homozygous sickle cell (HbSS) or sickle beta-zero-thalassemia (HbS/β0), as confirmed by high performance liquid chromatography or haemoglobin electrophoresis.
2. Body weight ≥5 kg at the time of screening.
3. If treated with an anti-sickling agent such as hydroxyurea, the weight-adjusted dose must be stable for 3 months before screening/enrolment.
4. Provision of signed and dated written informed consent from parents/legal guardians prior to any study specific procedures not part of standard medical care.

Exclusion criteria

1. History of transient ischaemic attack or cerebrovascular event/accident (ischaemic or haemorrhagic), severe head trauma, intracranial haemorrhage, intracranial neoplasm, arteriovenous malformation, aneurysm, or proliferative retinopathy.
2. Significantly underdeveloped with regards to height, weight or head circumference for age, as judged by the Investigator.
3. Severe developmental delay (eg, cerebral palsy or mental retardation).
4. Receiving chronic treatment (>3 days/week) with non-steroidal anti-inflammatory drugs (NSAIDs).
5. Receiving chronic treatment with anticoagulants or antiplatelet drugs that cannot be discontinued.
6. Moderate or severe hepatic impairment, defined as laboratory values of alanine aminotransferase (ALT) >2 × upper limit of normal (ULN), total bilirubin >2 × ULN (unless judged by the Investigator to be caused by haemolysis), albumin <35 g/L and international normalised ratio (INR) >1.4, or symptoms of liver disease (eg, ascites).
7. Renal failure requiring dialysis.
8. Active pathological bleeding or increased risk of bleeding complications according to the Investigator.
9. Haemoglobin <6 g/dL from test performed at Screening (Visit 1).
10. Platelets <100 × 10^9/L from test performed at Screening (Visit 1).
11. Patient considered to be at risk of bradycardic events (eg, known sick sinus syndrome or second or third degree atrioventricular block).
12. Concomitant oral or intravenous therapy with moderate or strong CYP3A4 inhibitors, CYP3A4 substrates with narrow therapeutic indices, or strong CYP3A4 inducers that have not been stopped at least 5 half-lives before dose administration.
13. Patient breastfed by mother who is under treatment of strong CYP3A4 inhibitors,
14. Active untreated malaria. Patients with suspected malaria at Screening (Visit 1) will be tested.
15. Surgical procedure planned to occur during the study including 5 days after ticagrelor administration.
16. Known hypersensitivity or contraindication to ticagrelor.
17. Concern for the inability of the patient or parents to comply with study procedures and/or follow-up.
18. Any condition which, in the opinion of the Investigator, would make it unsafe or unsuitable for the patient to participate in this study.
19. Previously administered ticagrelor in the present study.
20. Participation in another clinical study with an investigational medicinal product (IMP) or device during the last 30 days preceding screening/enrolment.
21. Involvement of member of patient's family in planning and/or conduct of the study (applies to both AstraZeneca personnel and personnel at study centre).

Ages: 1 Day to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Ticagrelor | 1,2,4,6 hours post dose
  This measure is obtained from observed plasma concentrations
Area under plasma concentration curve | 1,2,4,6 hours post dose
  This measure is obtained from the population PK analysis
CL/F (Oral clearance) | 1,2,4,6 hours post dose
  This measure is obtained from the population PK analysis.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) for active metabolite (AR-C124910XX) | 1,2,4,6 hours post dose
Area under plasma concentration curve | 1,2,4,6 hours post dose
Assessment of ticagrelor suspension for palatability | Day 1, single timepoint assessment
  Questionnaire with one five-options question reflecting different degrees of patients willingness to swallow, from "swallowed without problem" to "vomited up medication".

CONTACTS AND LOCATIONS:
Locations (8):
- Research Site, Edegem, Belgium
- Research Site, Genova, Italy
- Kenya (2):
  - Research Site, Kisumu
  - Research Site, Nairobi
- Lebanon (2):
  - Research Site, Beirut
  - Research Site, Tripoli
- Research Site, Madrid, Spain
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Duniva Inusa BP, Inati A, Maes P, Githanga J, Ogutu B, Abboud MR, Miano M, Cela E, Nduba V, Niazi M, Astrand M, Persson K, Berggren A, Carlson G. Pharmacokinetics and safety of ticagrelor in infants and toddlers with sickle cell disease aged <24 months. Pediatr Blood Cancer. 2021 May;68(5):e28977. doi: 10.1002/pbc.28977. Epub 2021 Feb 25. PMID 33629819
- See also: Study results information posted to AstraZeneca Cinical Trials Webiste — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/View?id=25368